CLINICAL TRIAL: NCT03778879
Title: A Phase 1b Trial of Neoadjuvant Stereotactic Body Radiotherapy With or Without CCR2 Inhibitor (CCX872-B) Immunotherapy for Preoperative Treatment of Resectable Pancreatic Cancer
Brief Title: Pre-operative Stereotactic Body Radiation Therapy for Pancreatic Adenocarcinoma With or Without CCX872-B
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: CCX872-B will not be available in sufficient quantity to conduct the study.
Sponsor: Alan Katz (Other)
Responsible Party: Sponsor-Investigator, Alan Katz, Associate Professor, University of Rochester
Organization: University of Rochester (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UGIP18131
Record Dates: First submitted 2018-12-15; First posted 2018-12-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Adenocarcinoma of the Pancreas; Pancreas Cancer
Keywords: Adenocarcinoma; Pancreas; Radiation Therapy; CCX872-B
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1:With CCX872-B (Experimental): Concurrent SBRT 25 Gy in 5 fractions over 5-7 days, and 21 days of CCX872-B therapy. CCX872-B 150 mg by mouth twice daily approximately 12 hours apart.
  Interventions: Drug: CCX872-B
- Group 2:Without CCX872-B (No Intervention): SBRT Alone: 25 Gy in 5 fractions over 5-7 days

INTERVENTIONS:
Drug: CCX872-B — CCX872-B concurrent with stereotactic body radiation therapy for pancreatic adenocarcinoma.
  Arms: Group 1:With CCX872-B

SUMMARY:
Standard treatment for newly diagnosed operable pancreatic cancer usually involves undergoing surgery first and then receiving chemotherapy with or without radiation therapy. However, the pancreatic cancer often comes back after this treatment. Therefore, the investigators are studying whether giving treatment prior to surgery can help decrease the risk the cancer returns.

Stereotactic Body Radiation Therapy (SBRT) is a highly focused type of radiation therapy commonly used in the treatment of pancreatic cancer. This treatment has been shown to be safe and effective for the preoperative treatment of pancreatic cancer. The purpose of this study is to determine if combining an experimental drug, CCX872-B, with SBRT continues to be safe and whether the combination treatment may be more effective at boosting the participant's immune system's ability to kill the pancreatic cancer.

DETAILED DESCRIPTION:
The investigators have shown that preoperative SBRT followed by surgical resection is feasible and safe in patients in the previous trial UGIP14107. The investigators have also presented preclinical evidence that inhibiting entry of CCR2+ IM using a small molecule antagonist against CCR2 results in enhanced efficacy of RT 26. The investigators hypothesize that inhibition of the CCR2 axis can potentially up regulate the immune response following radiation, therefore leading to a more robust tumor killing response. In preclinical studies, CCR2 inhibitor has little effect in the absence of RT, therefore, the investigators are not including a drug therapy alone group. To test this hypothesis, a phase Ib clinical trial has been proposed to evaluate the effect of combining stereotactic body radiotherapy with CCR2 inhibition in the neoadjuvant treatment of surgically resectable adenocarcinoma of the head of the pancreas.

The study will consist of two parts in sequential fashion. The first fifteen patients will be assigned to Group 1 and undergo SBRT with CCR2 inhibitor CCX872-B. The primary objective is to establish safety and feasibility of the treatment and analyze biomarkers to determine if combined treatment can stimulate an immune response in human patients. A second group of 5 patients will undergo SBRT alone as a comparison group for biomarker immune response.

The investigators would like to proceed with SBRT and CCX872-B as Group 1 given the investigators already have sufficient data from UGIP14107 to show that SBRT is safe and feasible and studying the combination of SBRT with CCX872-B is the primary scientific objective of this study. If unexpected safety issues occur with Group 1, the investigators would consider closing trial at that time without enrolling any patients in Group 2 which would reduce the number of patients exposed to the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with pathologically proven diagnosis of adenocarcinoma of the head of the pancreas
2. CT w/ contrast or MRI of the abdomen and pelvis with contrast within 6 weeks prior to registration
3. CT chest or PET/CT within 6 weeks prior to registration
4. Clinically determined to be resectable based on NCCN Criteria 3.2017: No arterial tumor contact (celiac axis, superior mesenteric artery or common hepatic artery) and no tumor contact with the superior mesenteric vein or portal vein, or < 180 degrees contact without vein contour irregularity
5. No evidence of metastatic disease and/or non-regional lymph node metastases
6. Adequate cardiopulmonary reserves to tolerate surgery
7. ECOG performance status 0-2
8. Adequate bone marrow function defined as follows: White blood cell> 3000cells/mm^3, Absolute neutrophil count (ANC) ≥ 1500 cells/mm3, Platelets ≥ 100,000 cells/mm3, Hemoglobin ≥ 9.0 g/dl
9. Male or female subjects, aged at least 18 years; Female subjects of childbearing potential may participate if adequate contraception is used during, and for at least the three months after study completion; Male subjects with partners of childbearing potential may participate in the study if they had a vasectomy at least 6 months prior to randomization or if adequate contraception is used during, and for at least the three months after study completion; Adequate contraception is defined as resulting in a failure rate of less than 1% per year
10. Patient must sign study specific informed consent prior to study entry
11. Anticipated life expectancy ≥ 12 weeks; -

Exclusion Criteria:

1. Prior surgical resection of any pancreatic malignancy
2. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years
3. Any prior systemic or radiation treatment, including investigational treatments, of the patient's pancreatic tumor.
4. Prior radiotherapy to the region of pancreatic cancer that would result in overlap of radiation therapy fields
5. Severe, active comorbidity, defined as follows:

   1. Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
   2. Transmural myocardial infarction within the last 6 months
   3. Clinically significant ECG abnormalities e.g. QTcF >450msec
   4. Acute viral, bacterial or fungal infection requiring intravenous antibiotics at the within 4 weeks of registration
   5. Known active HIV, HBV or HCV infections
   6. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days prior to registration.
   7. Uncontrolled diabetes or hypertension
   8. Serious psychiatric illness or altered mental status
6. Severe, uncorrectable hepatic insufficiency and/or coagulation defects due to liver failure
7. Any evidence of distant metastases (M1)
8. (ONLY applies for Group 1 patients taking CCX872-B )Taking agents known to be strong inhibitors or inducers of CYP3A4 or UGT1A1 within 2 weeks prior to Day 1 dosing; these include atazanavir, boceprevir, clarithromycin, conivaptan, gemfibrozil, grapefruit juice, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir, mibefradil, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, voriconazole, rifampin, and carbamazepine; use of these drugs must be avoided during the study and until 2 weeks after stopping CCX872-B treatment -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who complete radiation therapy, drug treatment and surgery | 6 weeks
  Number of patients who proceed through radiation and drug treatment and undergo surgical resection in a timely manner.
Percentage of patients who are ineligible for surgical resection due to toxicity from SBRT + CCX872-B or SBRT alone | 12 weeks
  Assessment of whether patients are made ineligible for surgical resection solely due to toxicities from SBRT + CCX872-B or SBRT alone.
  Measure of Grade 3 toxicity directly attributable to SBRT+ CCX872-B or SBRT alone.
  Analyze rate of grade 2 or greater acute toxicity caused by SBRT with or without CCX872-B.
  Determination of intraoperative and postoperative surgical morbidity following neoadjuvant treatment including the amount of fibrosis and total operative time.

SECONDARY OUTCOMES:
Number of participants with no further growth of cancer at original site | 2 years
  Count subjects with no further growth of cancer at original site
Number of subjects with recurrence of cancer in other body sites | 2 years
  Compare recurrence locations (metastases to other organs or non-regional adenopathy) of treated patients relative to historical controls
Mean time to progression of pancreatic cancer | 4 years
  Duration of progression free survival of treated patients
Mean time to death | 4 years
  Measure duration of survival of treated patients

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No